CLINICAL TRIAL: NCT04898114
Title: Effectiveness of Nebulized Magnesium Sulfate Combined With Sildenafil Citrate in Persistent Pulmonary Hypertension of Newborn
Brief Title: Nebulized Magnesium Sulfate and Sildenafil for Persistent Pulmonary Hypertension of Newborn
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elsayed Abdelkreem, Lecturer of Pediatrics, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neb-Mag-2
Record Dates: First submitted 2021-05-20; First posted 2021-05-24 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Persistent Pulmonary Hypertension of Newborn
Keywords: neonate; persistent fetal circulation; persistent pulmonary hypertension of the newborn; PPHN; Magnesium Sulfate; Nebulizer; hypoxia; mechanical ventilation
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome; Hypoxia | interventions — Magnesium Sulfate; Sildenafil Citrate; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Two groups of neonates with PPHN on mechanical ventilation: (1) NebMag group: receive nebulized magnesium sulfate and oral sildenafil citrate; (2) Control group: receive nebulized placebo (isotonic saline) and oral sildenafil citrate.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each neonate will be assigned a unique identification number. Pharmacy will fill the active and placebo preparations in similar containers with sealed code for identification. Participants' families, treating clinicians, nurses, echocardiographers, and data collectors will be unaware of group assignment and drug/placebo therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NebMag (Experimental): Nebulized magnesium sulfate and oral sildenafil
  Interventions: Drug: Magnesium sulfate; Drug: Sildenafil Citrate
- Control (Placebo Comparator): Nebulized placebo (isotonic saline) and oral sildenafil
  Interventions: Drug: Sildenafil Citrate; Other: Isotonic saline

INTERVENTIONS:
Drug: Magnesium sulfate — Nebulized magnesium sulfate (4 ml of 6.4% solution) every 15 minutes
  Other Names: MgSO4
  Arms: NebMag
Drug: Sildenafil Citrate — Oral sildenafil citrate at an initial dose of 1 mg/kg, with incremental increases by 0.5 mg/kg every 6 hours till reaching a target dose of 2mg/kg every 6 hours.
  Other Names: Viagra
Other: Isotonic saline — Nebulized isotonic saline (4 ml) every 15 minutes
  Other Names: 0.9% NaCl
  Arms: Control

SUMMARY:
The aim of this study is to evaluate the effectiveness of nebulized magnesium sulfate combined with sildenafil citrate, compared with sildenafil citrate alone, in treating neonates with severe persistent pulmonary hypertension on mechanical ventilation.

DETAILED DESCRIPTION:
Persistent pulmonary hypertension of newborn (PPHN) is a serious condition that results from failure of the normal postnatal circulatory transition and is associated with significant mortality and morbidity. Advanced medical treatment, such as inhaled nitric oxide (iNO), high-frequency ventilation (HFV), and extracorporeal membrane oxygenation (ECMO) are commonly not available in developing countries. Intravenous magnesium sulfate has been shown to alleviate pulmonary hypertension but is associated with systemic hypotension and is less effective compared with iNO and sildenafil. Nebulized magnesium sulfate has been reported to be more effective and safer compared with intravenous magnesium sulfate in treating neonates with PPHN on mechanical ventilation. Combined nebulized magnesium and sildenafil has been studied in a small trial on spontaneously breathing neonates with PPHN but not on those connected to mechanical ventilation.

The aim of this study is to evaluate the effectiveness of nebulized magnesium sulfate combined with sildenafil citrate, compared with sildenafil citrate alone, in treating neonates with severe PPHN on mechanical ventilation. We hypothesize that neonates with severe PPHN connected to mechanical ventilation could benefit from taking continuous nebulization of magnesium sulfate combined besides sildenafil.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 36 weeks
* Birth weight between 2.5 and 4 kg.
* Post-natal age between 6 and 72 hours.
* PPHN confirmed by echocardiography
* Oxygenation index (OI) > 30 on two occasions at least 15 minutes apart
* Connected to Mechanical Ventilation

Exclusion Criteria:

* Failure to obtain informed consent
* Newborns to mothers who received magnesium sulfate within 48 hours before labor.
* Congenital heart diseases, other than patent ductus arteriosus and foramen ovale.
* Major congenital anomalies (including congenital diaphragmatic hernia and lung hypoplasia).
* Prior need for cardiopulmonary resuscitation.
* Mean arterial blood pressure (MABP) < 35 mmHg despite therapy with volume infusions and vasoactive inotropes.
* Impaired kidney function.
* Prior administration of pulmonary vasodilators.
* Gastrointestinal intolerance or bleeding

Ages: 6 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Oxygenation index (OI) | From baseline to 2, 6, 12, and 24 hours following study drug administration
  OI will be calculated using the following formula: OI = [(FiO2 × MAP) / PaO2] (FiO2, fraction of inspired oxygen expressed in %; MAP, mean airway pressure in cmH2O/mmHg; and PaO2, partial pressure of arterial oxygen in mmHg).

SECONDARY OUTCOMES:
Change in Mean arterial blood pressure (MABP) | From baseline to 2, 6, 12, and 24 hours following study drug administration.
Change in Vasoactive Inotropic Score (VIS) | From baseline to 2, 6, 12, and 24 hours following study drug administration.
  The VIS will be calculated using the following formula: VIS = dopamine dose (µg/kg/min) + dobutamine dose (µg/kg/min) + 100 × epinephrine dose (µg/kg/min) + 100 × norepinephrine dose (µg/kg/min) + 10 × milrinone dose (µg/kg/min) + 10,000 × vasopressin dose (U/kg/min).
Change in Pulmonary artery systolic pressure (PASP) | From baseline to 24 hours after study drug administration
  PASP will be estimated by echocardiography using the modified Bernoulli equation: PASP = (TRJV2 × 4) + RAP (TRJV, tricuspid regurgitation jet velocity; RAP, right atrial pressure).
Change in Serum magnesium level | From baseline to 24 hours after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Elsayed Abdelkreem, MD, PhD, Principal Investigator — Sohag University
Locations (1):
- Neonatal Intensive Care Unit, Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual participant data will be available from the principal investigator upon reasonable request
Supporting Information: Study Protocol
Time Frame: Three years after publication of the study results
Access Criteria: Unidentified individual participant data can be requested from the principal investigator

REFERENCES:
- [Background] Abdelkreem E, Mahmoud SM, Aboelez MO, Abd El Aal M. Nebulized Magnesium Sulfate for Treatment of Persistent Pulmonary Hypertension of Newborn: A Pilot Randomized Controlled Trial. Indian J Pediatr. 2021 Aug;88(8):771-777. doi: 10.1007/s12098-020-03643-y. Epub 2021 Jan 8. PMID 33415555
- [Background] Mandell E, Kinsella JP, Abman SH. Persistent pulmonary hypertension of the newborn. Pediatr Pulmonol. 2021 Mar;56(3):661-669. doi: 10.1002/ppul.25073. PMID 32930508
- [Background] El-Khuffash A, McNamara PJ, Breatnach C, Bussmann N, Smith A, Feeney O, Tully E, Griffin J, de Boode WP, Cleary B, Franklin O, Dempsey E. The use of milrinone in neonates with persistent pulmonary hypertension of the newborn - a randomised controlled trial pilot study (MINT 1): study protocol and review of literature. Matern Health Neonatol Perinatol. 2018 Dec 3;4:24. doi: 10.1186/s40748-018-0093-1. eCollection 2018. PMID 30524749
- [Background] Lai MY, Chu SM, Lakshminrusimha S, Lin HC. Beyond the inhaled nitric oxide in persistent pulmonary hypertension of the newborn. Pediatr Neonatol. 2018 Feb;59(1):15-23. doi: 10.1016/j.pedneo.2016.09.011. Epub 2017 Aug 10. PMID 28923474
- [Background] Nakwan N. The Practical Challenges of Diagnosis and Treatment Options in Persistent Pulmonary Hypertension of the Newborn: A Developing Country's Perspective. Am J Perinatol. 2018 Dec;35(14):1366-1375. doi: 10.1055/s-0038-1660462. Epub 2018 Jun 19. PMID 29920641
- [Background] He Z, Zhu S, Zhou K, Jin Y, He L, Xu W, Lao C, Liu G, Han S. Sildenafil for pulmonary hypertension in neonates: An updated systematic review and meta-analysis. Pediatr Pulmonol. 2021 Aug;56(8):2399-2412. doi: 10.1002/ppul.25444. Epub 2021 May 13. PMID 33983650
- [Background] Ho JJ, Rasa G. Magnesium sulfate for persistent pulmonary hypertension of the newborn. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD005588. doi: 10.1002/14651858.CD005588.pub2. PMID 17636807